CLINICAL TRIAL: NCT06967311
Title: Microbial and Human Determinants of the Onset of IBD Flares
Brief Title: Human and Microbial Determinants of the Onset of IBD Flares
Status: Recruiting | Type: Observational
Sponsor: Viome (Industry)
Collaborators: Universidade Federal de Santa Catarina (Other)
Responsible Party: Sponsor
Other Study IDs: V233
Record Dates: First submitted 2025-03-28; First posted 2025-05-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: IBD (Inflammatory Bowel Disease)
Keywords: observational; IBD; microbiome
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect and retain whole blood, dried blood spots, stool, and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease (IBD): Individuals diagnosed with IBD

SUMMARY:
This study will collect longitudinal biological samples and survey data to identify the triggers of IBD flares.

DETAILED DESCRIPTION:
This is a longitudinal observational study whose goals are to identify:

Microbial and human molecular triggers of IBD relapses, Microbial and human molecular pathways strongly associated with flares that could be targeted with nutrition with a therapeutic potential, Biomarkers of IBD for Dx purposes, Identify microbial functions associated with release of BH4.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Universidade Federal de Santa Catarina (UFSC) Hospital, under care of Dr. Vivian Menegassi

Exclusion Criteria:

* Cancer Diagnosis/Treatment
* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Crohn's Disease or Ulcerative Colitis that are patients at Universidade Federal de Santa Catarina (UFSC) Hospital and under care of Dr. Vivian Menegassi
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Stool microbial KEGG orthologs (KOs) associated with IBD | For 12 months from enrollment
  Metatranscriptomic tests will be used to quantify microbial KOs in stool samples. At the end of the study, we will use machine learning to identify KOs whose expression is associated with IBD.

CONTACTS AND LOCATIONS:
Locations (1):
- LABOX, Department of Biochemistry, Universidade Federal de Santa Catarina, Florianópolis, Santa Catarina, Brazil